CLINICAL TRIAL: NCT04710849
Title: Relationship Between Plasma Metabolome and the Efficacy of Systemic Glucocorticoid in Acute Exacerbation of Chronic Obstructive Pulmonary Disease
Brief Title: Relationship Between Plasma Metabolome and the Efficacy of Systemic Glucocorticoid in AECOPD
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, li qiuyu, Attending Doctor of Department of Respiratory and Critical Care Medicine, Peking University Third Hospital
Other Study IDs: PUTH-COPD001
Record Dates: First submitted 2021-01-10; First posted 2021-01-15 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2021-01

CONDITIONS: COPD; COPD Exacerbation Acute
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Treatment Failure Group: The diagnostic criteria of AECOPD is defined in global initiative for chronic obstructive lung disease (GOLD 2016). According to the efficacy of systemic hormone therapy during hospitalization, they were divided into treatment success group and treatment failure group. Definition of systemic glucocorticoid treatment failure during hospitalization is (Reference: Crisafulli E, Torres A, Huerta A, et al. COPD, 2016, 13(1): 82-92): The following occurs from the 2nd to the 7th day after admission Situation: ①Need to receive mechanical ventilation treatment or need to be admitted to the ICU due to illness; ②72 hours after the initial anti-infective treatment, clinical signs of infection persist and need to change antibiotic treatment; ③Death from any cause.
  Interventions: Diagnostic Test: Serum metabolic markers
- Treatment Success Group: The diagnostic criteria of AECOPD is defined in global initiative for chronic obstructive lung disease (GOLD 2016). According to the efficacy of systemic hormone therapy during hospitalization, they were divided into treatment success group and treatment failure group. The treatment success group was defined as not meeting any of the following conditions for failure of systemic hormone therapy during hospitalization (reference: Crisafulli E, Torres A, Huerta A, et al. COPD, 2016, 13(1): 82-92): ①Need to receive mechanical ventilation treatment or need to be admitted to the ICU due to illness; ②72 hours after the initial anti-infective treatment, clinical signs of infection persist and need to change antibiotic treatment; ③Death from any cause.
  Interventions: Diagnostic Test: Serum metabolic markers

INTERVENTIONS:
Diagnostic Test: Serum metabolic markers — Ultraperformance liquid chromatography / mass spectrometry (LC-MS) and gas chromatography / mass spectrometry (GC-MS) methods for analysis of the metabolites in AECOPD patients and compare the metabolites profiles between patients with systemic glucocorticoid treatment success and treatment failure.
  Other Names: Metbolomics

SUMMARY:
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) significantly increases the mortality of the patients with COPD. Guidelines have recommended systemic glucocorticoid as regular treatment. Recently, evidences have shown that systemic glucocorticoid cannot not be benefit to all of the patients with AECOPD. Thus the problem that how the clinicians can screen the patients who can benefit from systemic glucocorticoid needs to be solved urgently.

DETAILED DESCRIPTION:
Acute exacerbation of chronic obstructive pulmonary disease (AECOPD) significantly increases the mortality of the patients with COPD. Guidelines have recommended systemic glucocorticoid as regular treatment. Recently, evidences have shown that systemic glucocorticoid cannot not be benefit to all of the patients with AECOPD. Thus the problem that how the clinicians can screen the patients who can benefit from systemic glucocorticoid needs to be solved urgently. A previous study found that plasma metabolome changed significantly after dexamethasone treatment in health participants. Furthermore, inter-person variability was high and remained uninfluenced by treatment, suggesting the potential of metabolomics for predicting the efficacy and side effects of systemic glucocorticoid. Our previous study found that serum metabolites profile in COPD patients differed from that in controls. Therefore, the investigators hypothesized that metabolome changes in patients with AECOPD may be associated with the efficacy of systemic glucocorticoid. In this study, the investigators will utilize ultraperformance liquid chromatography / mass spectrometry (LC-MS) and gas chromatography / mass spectrometry (GC-MS) methods for analysis of the metabolites in AECOPD patients and compare the metabolites profiles between patients with systemic glucocorticoid treatment success and treatment failure. The investigators aim to detect the metabolic biomarkers and metabolic pathways which are related to efficacy of systemic glucocorticoid and contribute to the precise treatment of COPD.

ELIGIBILITY:
Inclusion Criteria:

* Patients who meet the diagnostic criteria for acute exacerbation of chronic obstructive pulmonary disease in GOLD 2016 and require hospitalization.

Exclusion Criteria:

* Bronchial asthma, bronchiectasis and other airflow obstructive diseases;
* Combined with community-acquired pneumonia, hospital-acquired pneumonia or aspiration pneumonia;
* Combined with severe liver and kidney insufficiency;
* Malignant tumor;
* Immune deficiency due to chemotherapy or HIV infection;
* Received systemic hormone therapy due to acute exacerbation of chronic obstructive pulmonary disease within 1 month before this admission;
* Severe trauma or stress, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A prospective study was conducted to recruit consecutive patients from January 1, 2020 to January 1, 2021 who were hospitalized in the Department of Respiratory and Critical Care Medicine in Peking University Third Hospital and met the diagnostic criteria of acute exacerbation of chronic obstructive pulmonary disease (AECOPD) in Global Initiative for Chronic Obstructive Lung Diseas 2016 (GOLD 2016).
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-02-01 (Estimated); Primary Completion 2024-02-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
Metabolic markers related to systemic glucocorticoid therapy | 1 year
  Through metabolomics research methods such as liquid chromatography-mass spectrometry and gas chromatography-mass spectrometry, study the metabolic marker group profile of patients with acute exacerbation of COPD before receiving systemic glucocorticoid therapy, and look for possible systemic metabolic markers related to the short-term and long-term effects of glucocorticoids.

SECONDARY OUTCOMES:
Length of hospital stay | 1 year
  The time interval from admission to discharge of the patient this time
Time from discharge to the next exacerbation | 1 year
  The time interval from the patient's discharge from the hospital to the next acute exacerbation of chronic obstructive pulmonary disease
Side effects of glucocorticoid therapy | 1 year
  Any side effects related to glucocorticoid therapy, including osteoporosis, hyperglycemia, infection, etc.
Mortality within 1 year | 1 year
  The mortality rate of the patients within 1 year after enrollment, including overall mortality and COPD-related mortality
Acute exacerbation frequency | 1 year
  The number of acute exacerbations of chronic obstructive pulmonary disease in the one year follow-up after enrollment
mMRC score | 1 year
  Evaluate the severity of dyspnea through a modified version of the British Medical Research Council Respiratory Questionnaire (mMRC)
CAT score | 1 year
  Evaluate the severity of dyspnea through the COPD assessment Test questionnaire (CAT)
Changes in pulmonary function | 1 year
  Ventilation function and changes indicated by the patient's pulmonary function test

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Li QY, An ZY, Pan ZH, Qi RY. Rationale and design of REGULATE: an observational study protocol for relationship between plasma metabolome and the efficacy of systemic glucocorticoid in acute exacerbation of chronic obstructive pulmonary disease. BMC Pulm Med. 2021 Jul 28;21(1):250. doi: 10.1186/s12890-021-01614-3. PMID 34320980